CLINICAL TRIAL: NCT05853900
Title: A Randomized Double-blind, Parallel-Group, Virtual Study to Evaluate the Effectiveness and Safety of Two Digital Therapeutics in Late Adolescents and Adults for the Prevention of Episodic Migraine
Brief Title: Study of Two Digital Therapeutics for the Prevention of Episodic Migraine
Acronym: ReMMi-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-132-R-001
Record Dates: First submitted 2023-04-18; First posted 2023-05-11 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Migraine; Episodic Migraine; Headache; Headache, Migraine
Keywords: Prescription digital therapeutic (PDT); Software as a Medical Device (SaMD); Smartphone app
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Arm A (Experimental): Mobile application A as a software-based intervention for the preventive treatment of episodic migraine in late adolescents and adults.
  Interventions: Device: ReMMi-D Digital Therapeutic
- Arm B (Experimental): Mobile application B is an investigational digital therapeutic that is being studied for the preventative treatment of episodic migraine.
  Interventions: Device: ReMMi-D Digital Therapeutic

INTERVENTIONS:
Device: ReMMi-D Digital Therapeutic — Evaluate the effectiveness and safety of prescription mobile applications that provide an interactive, software-based intervention for the preventative treatment of episodic migraine in late adults and adolescents.

SUMMARY:
Randomized study of two digital therapeutics for the prevention of episodic migraine

DETAILED DESCRIPTION:
The purpose of this randomized ReMMi-D trial is to evaluate the effectiveness and safety of two prescription mobile applications that provide an interactive, software-based intervention for the preventative treatment of episodic migraine in late adolescents and adults.

ELIGIBILITY:
Inclusion Criteria:

* A participant will be eligible for entry into the study if all of the following criteria are met:

  1. Willing and able to provide written informed consent to participate in the study, attend study visits, and comply with study-related requirements and assessments.
  2. Lives in the United States.
  3. Adult or late adolescent, 18 years of age or older at the time of informed consent.
  4. Fluent in written and spoken English, confirmed by ability to read and understand the informed consent form.
  5. The following will be physician-reviewed: Participant has at least a 1-year history of migraine (with or without aura) consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition.

     1. Age of onset of migraines prior to 50 years of age
     2. Migraine attacks, on average, lasting 4-72 hours if untreated
     3. Per participant report, 4-14 migraine days per month within the last 3 months prior to the Screening Visit (a month is defined as 28 days)
     4. Four to fourteen migraine days during the run-in period
  6. Is currently managing migraines with ≥1 prescription acute treatment and/or prescription first or second-line preventive medications, as assessed by a physician.
  7. Is the sole user of an iPhone with an iPhone operating system (iOS) 14 or later or a smartphone with an Android operating system (OS) 11 or later and is willing to download and use the Study App required by the protocol.
  8. Is willing and able to receive SMS text messages and push messages on their smartphone.
  9. Is the owner of, and has regular access to, an email address.
  10. Has regular access to the Internet via cellular data plan and/or wifi.

Exclusion Criteria:

* A participant will not be eligible for study entry if any of the following criteria are met:

  1. History of basilar migraine or hemiplegic migraine.
  2. Active chronic pain syndromes, such as fibromyalgia, chronic pelvic pain, or complex regional pain syndrome (CRPS).
  3. Other pain syndromes (including trigeminal neuralgia), psychiatric conditions (such as major depressive episode, bipolar disorder, major depressive disorder, schizophrenia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, might interfere with study assessments.
  4. History of, treatment for, or evidence of, alcohol or drug abuse within the past 12 months (48 weeks) or having met DSM-V criteria for any significant substance use disorder within the past 12 months (48 weeks) from the date of the screening visit.
  5. History of use of analgesics (e.g., nonsteroidal anti-inflammatory drugs [NSAIDs] or acetaminophen, including opioids) or butalbital on ≥ 15 days per month during the 3 months (12 weeks) prior to the Screening Visit or during the run-in period.
  6. Currently taking a prescription anti-calcitonin gene-related peptide (CGRP) for either episodic or chronic migraine.
  7. Post-traumatic headache, persistent post-traumatic headache, or post-concussion syndrome.
  8. Other significant episodic or chronic medical condition(s) that in the opinion of the Investigator, may confound the interpretation of findings to inform PDT development.
  9. Failure to adhere with or inability to complete Study App inputs and onboarding activities during the run-in period. Participants who are not adherent during the run-in period are not eligible for study entry.
  10. Previous enrollment in any digital therapeutics pilot or pivotal study for a migraine indication.
  11. Participation in any other investigational clinical study while participating in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, Principal Investigator — ObvioHealth
Locations (1):
- Click Therapeutics, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (CT-132): Mobile application A as a software-based intervention for the preventive treatment of episodic migraine in late adolescents and adults.
- Arm B (Digital Control): Mobile application B is an investigational digital therapeutic that is being studied for the preventative treatment of episodic migraine.
Period: Overall Study
Arm/Group | Arm A (CT-132) | Arm B (Digital Control)
Started | 285 | 283
Completed | 255 | 262
Not Completed | 30 | 21

BASELINE CHARACTERISTICS:
Groups:
- Arm A (CT-132): Mobile application A (CT-132) as a software-based intervention for the preventive treatment of episodic migraine in late adolescents and adults.
- Arm B (Digital Control): Mobile application B (Digital Control) is an investigational digital therapeutic that is being studied for the preventative treatment of episodic migraine.
- Total: Total of all reporting groups
Arm/Group | Arm A (CT-132) | Arm B (Digital Control) | Total
Number analyzed (Participants) | 285 | 283 | 568
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (10.4) | 38.9 (10.3) | 38.7 (10.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 263 | 265 | 528
  Male | 12 | 13 | 25
  Other | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 13 | 23
  Not Hispanic or Latino | 275 | 270 | 545
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 269 | 261 | 530
  More than one race | 8 | 12 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 285 | 283 | 568

OUTCOME MEASURES:

1. Primary Outcome: Change in MMD (Monthly Migraine Days)
Description: Change in the number of MMDs from baseline (28-day Run-in Period) to Week 12 (previous 28 days, Week 9 through Week 12).
Time Frame: Baseline (28-day Run-in Period) to Week 12 (previous 28 days, Week 9 through Week 12)
Population: Intent-to-treat Population, all enrolled participants who were randomized, based on the assigned intervention in the randomization and recorded in the database.
Measure: Least Squares Mean (95% Confidence Interval); unit: migraine days per month
Arm/Group | Arm A (CT-132) | Arm B (Digital Control)
Number analyzed (Participants) | 266 | 264
migraine days per month | -3.04 [-3.49 to -2.58] | -2.14 [-2.59 to -1.69]

2. Secondary Outcome: Participants Who Have at Least a 50% Reduction From Baseline
Description: Participants who have at least a 50% reduction from baseline (28-day Run-in Period) in the number of MMDs to Week 12 (previous 28 days, Week 9 through Week 12)
Time Frame: Baseline (28-day Run-in Period) to Week 12 (previous 28 days, Week 9 through Week 12)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (CT-132) | Arm B (Digital Control)
Number analyzed (Participants) | 266 | 264
Participants
  Responder | 141 | 113
  Non-responder | 125 | 151

3. Secondary Outcome: Change From Baseline in the Number of MMD Recorded Over the Previous 28 Days at Week 4 and Week 8
Description: Change from baseline (28-day Run-in Period) in the number of MMDs recorded over the previous 28 days at Week 4 and at Week 8
Time Frame: Baseline (28-day Run-in Period) to Weeks 4 and 8
Population: The overall number of participant analyzed present the number of participant with data at the time interval the assessment was complete (at week 4 and at week 8).
Measure: Mean (Standard Deviation); unit: migraine days per month
Arm/Group | Arm A (CT-132) | Arm B (Digital Control)
Number analyzed (Participants) | 285 | 283
migraine days per month
  Change from Baseline at Week 4: number analyzed (Participants) | 280 | 278
  Change from Baseline at Week 4 | -1.58 (3.55) | -1.20 (3.31)
  Change from Baseline at Week 8: number analyzed (Participants) | 277 | 275
  Change from Baseline at Week 8 | -2.24 (3.92) | -1.87 (3.65)

4. Secondary Outcome: Change From Baseline in the Mean Number of MMD Over 12 Weeks
Description: Change from baseline (28-day Run-in Period) in the mean number of MMDs over 12 weeks.
Time Frame: Baseline (28-day Run-in Period) to Week 12
Measure: Mean (Standard Deviation); unit: migraine days per month
Arm/Group | Arm A (CT-132) | Arm B (Digital Control)
Number analyzed (Participants) | 266 | 264
migraine days per month | -3.35 (3.63) | -2.26 (3.67)

5. Secondary Outcome: Change in Number of Headaches With at Least Moderate Severity From Baseline to Week 12
Description: Change in the number of headaches with at least moderate severity from baseline (28-day run-in period) to Week 12 (previous 28 days, Week 9 through Week 12).
Time Frame: Baseline (28-day Run-in Period) to Week 12 (previous 28 days, Week 9 through Week 12)
Measure: Mean (Standard Deviation); unit: headaches
Arm/Group | Arm A (CT-132) | Arm B (Digital Control)
Number analyzed (Participants) | 266 | 264
headaches | -3.48 (2.66) | -2.87 (2.64)

6. Secondary Outcome: Change From Baseline in the Migraine-Specific Quality-of-Life Questionnaire v2.1 (MSQ) Total Score Over the Previous 28 Days at Week 4, Week 8, and Week 12
Description: Change from baseline in the Migraine-Specific Quality-of-Life Questionnaire v2.1 (MSQ) at Week 4, Week 8, and Week 12 The MSQ is a self-administered, 14-item instrument that is completed at baseline, Week 4, Week 8, and Week 12. Participants respond to items using a 6-point scale: "none of the time," "a little bit of the time," "some of the time," "a good bit of the time," "most of the time," and "all of the time," which are assigned scores of 1 to 6, respectively. Next, raw dimension scores are computed as a sum of recoded item scores and rescaled from a 0 to 100 scale such that higher scores indicate better quality of life.
Time Frame: Baseline (28-day Run-in Period) to Weeks 4, 8 and 12.
Population: The overall number of participant analyzed present the number of participant with data at the time-interval the assessment was complete (at week 4, at week 8 and at week 12).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (CT-132) | Arm B (Digital Control)
Number analyzed (Participants) | 284 | 283
score on a scale
  Change from Baseline to Week 4: number analyzed (Participants) | 251 | 249
  Change from Baseline to Week 4 | 6.16 (13.48) | 2.12 (13.42)
  Change from Baseline to Week 8: number analyzed (Participants) | 251 | 246
  Change from Baseline to Week 8 | 9.13 (15.82) | 4.30 (13.85)
  Change from Baseline to Week 12: number analyzed (Participants) | 254 | 261
  Change from Baseline to Week 12 | 11.95 (15.52) | 5.03 (16.26)

7. Secondary Outcome: Change From Baseline (28-day Run-in Period) in the Migraine Disability Assessment (MIDAS) to Week 12 (Previous 28 Days, Week 9 Through Week 12)
Description: Change from baseline in the Migraine Disability Assessment (MIDAS) at Week 4, Week 8, and Week 12 The Migraine Disability Assessment (MIDAS) questionnaire is a brief, self report 5-item questionnaire (scale: 0 - 90 for each of 5 subscales) designed to quantify headache-related disability over a 3-month period. The 5 subscale scores are summed to compute the MIDAS total score (scale: 0 - 450). Lower scores indicate less headache-related disability.
Time Frame: Baseline to Weeks 4, 8, and 12
Population: The overall number of participant analyzed present the number of participant with data at the time interval the assessment was complete (at week 4, at week 8, and at week 12).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (CT-132) | Arm B (Digital Control)
Number analyzed (Participants) | 285 | 283
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 251 | 251
  Change from Baseline at Week 4 | -5.27 (29.89) | -0.89 (30.31)
  Change from Baseline at Week 8: number analyzed (Participants) | 251 | 247
  Change from Baseline at Week 8 | -7.50 (31.14) | -0.85 (33.27)
  Change from Baseline at Week 12: number analyzed (Participants) | 255 | 262
  Change from Baseline at Week 12 | -10.55 (33.03) | -3.30 (29.52)

8. Secondary Outcome: Change From Baseline (28-day Run-in Period) to Week 12 (Previous 28 Days, Week 9 Through Week 12) in the Number of Migraines With Use of an Acute Migraine Medication
Description: Change in the number of migraines with use of an acute migraine medications from the run-in period to Weeks 9-12.
  The number of migraines with use of an acute medication will be counted for the run-in period and for post randomization period. The change from baseline will be calculated as number of migraines in weeks 9-12 minus number of migraines in the run-in period with use of an acute medication.
Time Frame: Baseline (28-day Run-in Period) to Week 12 (previous 28 days, Week 9 through Week 12)
Measure: Mean (Standard Deviation); unit: migraine
Groups:
- Arm A (CT-132): Mobile application A as a software-based intervention for the preventive treatment of episodic migraine in late adolescents and adults.
  ReMMi-D Digital Therapeutic: Evaluate the effectiveness and safety of prescription mobile applications that provide an interactive, software-based intervention for the preventative treatment of episodic migraine in late adults and adolescents.
- Arm B (Digital Control): Mobile application B is an investigational digital therapeutic that is being studied for the preventative treatment of episodic migraine.
  ReMMi-D Digital Therapeutic: Evaluate the effectiveness and safety of prescription mobile applications that provide an interactive, software-based intervention for the preventative treatment of episodic migraine in late adults and adolescents.
Arm/Group | Arm A (CT-132) | Arm B (Digital Control)
Number analyzed (Participants) | 266 | 264
migraine | -2.70 (2.38) | -2.50 (2.42)

9. Secondary Outcome: Change in the Number of Monthly Headache Days (MHDs) From Baseline to Week 12
Description: Change in the number of monthly headache days from baseline to Weeks 9-12
Time Frame: Baseline (28-day Run-in Period) to Week 12 (previous 28 days, Week 9 through Week 12)
Measure: Mean (Standard Deviation); unit: headache days per month
Arm/Group | Arm A (CT-132) | Arm B (Digital Control)
Number analyzed (Participants) | 266 | 264
headache days per month | -4.86 (4.29) | -3.69 (4.08)

ADVERSE EVENTS:
Time Frame: Baseline (28-day run-in period) through Week 12 (up to 16 weeks).
Description: Safety population included all randomized participants who were exposed to the study intervention (completed at least one task).
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/278 | 0/278
Serious Adverse Events (participants affected / at risk) | 1/278 | 0/278
Other Adverse Events (participants affected / at risk) | 22/278 | 16/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=278) | Arm B (N=278)
peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=278) | Arm B (N=278)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Procedural pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Infections and infestations) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Status migrainosus (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT05853900/Prot_001.pdf
  • Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT05853900/SAP_002.pdf